CLINICAL TRIAL: NCT05280301
Title: Assessment of Sous Vide Water Baths for Acute Rewarming of Frostbitten Extremities
Brief Title: Multicenter Sous Vide Frostbite
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Nicholas Daniel, DO, Assistant Professor, Dartmouth-Hitchcock Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY02001452
Record Dates: First submitted 2022-03-02; First posted 2022-03-15 (Actual); Results first posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Frostbite; Frostbite of Hand; Frostbite of Foot
MeSH Terms: conditions — Frostbite

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Sous vide device (Experimental): The intervention will be the use of a sous vide device to heat the water bath to 38 degrees celsius, rather than the traditional methods of manual water exchanges or placing the frostbitten tissue under running water.
  Interventions: Device: Sous Vide Device (SVD)

INTERVENTIONS:
Device: Sous Vide Device (SVD) — A basin will be filled to the marked line with water from jugs at room temperature, for each frozen extremity. The sous vide device (SVD) will be attached to the distal edge of the basin. The SVD will be turned on and set to maintain the bath at a constant 38 degrees celsius for 30 minutes duration. The thermometers will be powered on continuously and the researcher will record temperatures simultaneously from each thermometer and the SVD every 2 minutes. At the end of the 30 minute treatment, the extremity assessed by the researcher for warmth and pliability. If the extremity still feels cold or frozen, an additional 30 minutes in the water bath will commence, with subsequent reassessment. Rewarming will be considered complete when the affected tissue becomes red or purple, soft, and pliable.

SUMMARY:
The purpose of this study is to determine the efficacy of using sous vide devices for heating and maintaining the circulating warm water bath used in the rewarming of acute frostbite.

DETAILED DESCRIPTION:
Frostbite can be a devastating and limb threatening injury. Treatment involves active rewarming in a warm water bath at a consistent temperature, but maintaining the correct temperature water is clinically challenging. Currently these water baths are created and monitored manually - leading to poor rewarming and inefficient use of resources. The "sous vide" device offers an alternative to the manual water bath method. The specific aim of our study is to evaluate the safety, efficacy, and feasibility of use of the sous vide device in patients with extremity frostbite in a multicenter prospective cohort. Data demonstrating the ability of the sous vide device to warm and precisely maintain water bath target temperatures, in addition to expanded evidence of the safety of this modality, will support the broader use of sous vide devices in frostbite care.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or up
* Age <17 with parent or guardian consent
* Ability to understand English
* Ability to provide consent to the study
* Acute frostbite of the hands and/or feet

Exclusion Criteria:

* Children under age 18 without parent or guardian
* Frostbite that has already thawed
* Frostbite of tissue other than hands or feet
* Inability to understand English
* Inability to provide consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-11-25 (Actual); Study Completion 2024-11-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicholas Daniel, DO, Principal Investigator — Dartmouth-Hitchcock Medical Center
Locations (1):
- Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Sous Vide Rewarming Group: All patients with acute frostbite were approached for inclusion into the study group.
Period: Overall Study
Arm/Group | Sous Vide Rewarming Group
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Sous Vide Rewarming Group
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 6
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 6
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Rewarming
Description: Assess if frostbitten extremities can be thawed in a warm water bath created by the experimental device.
Time Frame: Up to 90 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Sous Vide Rewarming Group
Number analyzed (Participants) | 7
Participants | 7

2. Primary Outcome: Time to Rewarm in Minutes
Description: Measure the time required to rewarm frostbitten extremities until the extremity is reddish or purple in coloration, and soft and pliable
Time Frame: Up to 90 minutes
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | Sous Vide Rewarming Group
Number analyzed (Participants) | 7
Minutes | 10 [7 to 13]

3. Secondary Outcome: Ease of Use: Provider Review
Description: Providers will report ease of use of the rewarming modality by completing a survey. The survey consists of two questions requesting providers to indicate ease of use of the device on a scale from 0-10, where 0 indicates easy and 10 indicated difficult.
Time Frame: Immediately after rewarming, up to 90 minutes
Measure: Mean (Full Range); unit: score on a scale
Arm/Group | Sous Vide Rewarming Group
Number analyzed (Participants) | 7
score on a scale | 2.8 [1 to 7]

ADVERSE EVENTS:
Time Frame: Through the study completion, an average of 45 minutes.
Arm/Group | Sous Vide Rewarming Group
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-01-17): https://cdn.clinicaltrials.gov/large-docs/01/NCT05280301/Prot_SAP_001.pdf